CLINICAL TRIAL: NCT00437424
Title: A Pharmacokinetic Study of Brivanib (BMS-582664) in Subjects With Advanced Solid Tumor Malignancies and Normal Hepatic Function or Hepatocellular Carcinoma With Impaired Hepatic Function
Brief Title: A Study of Brivanib (BMS-582664) in Patients With Liver Cancer and Mild, Moderate or Severe Liver Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA182-015
Record Dates: First submitted 2007-02-14; First posted 2007-02-21 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2011-05

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Hepatocellular cancer; Other advanced solid malignancies
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — brivanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Brivanib

INTERVENTIONS:
Drug: Brivanib — Tablet, Oral, Brivanib 400 mg, based on Day 1 PK, QD, until progression
  Other Names: BMS-582664

SUMMARY:
The primary purpose of this protocol is to determine the effect of BMS-582664 on patients with hepatocellular carcinoma with varying levels of hepatic impairment

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a biopsy proven advanced solid tumor
* Subjects with a biopsy proven diagnosis of hepatocellular carcinoma conforming to child pugh classifications A, B, or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to determine the effect of BMS-582664 on subjects with varying levels of hepatic impairment and guide prescribers with regards to dosing in specialized populations | throughout the study

SECONDARY OUTCOMES:
To assess safety and tolerability of BMS-582664 in subjects with HCC with mild, moderate, and severe hepatic impairment and in subjects with advanced malignancies with normal hepatic function | by Day 1 and Day 28 Pharmacokinetics
To assess efficacy of BMS-582664 in subjects with advanced solid tumor malignancies and subjects with HCC by CT or MRI | every 6 weeks until disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- United States (4):
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - Usc/Norris Comprehensive Cancer Center, Los Angeles, California
  - Case Western Reserve University, Clleveland, Ohio
  - South Texas Accelerated Research Therapeutics, Llc, San Antonio, Texas
- Local Institution, Seville, Spain

REFERENCES:
- [Derived] El-Khoueiry A, Posey JA, Castillo Ferrando JR, Krishnamurthi SS, Syed S, Kollia G, Walters I, Fischer BS, Masson E. The effects of liver impairment on the pharmacokinetics of brivanib, a dual inhibitor of fibroblast growth factor receptor and vascular endothelial growth factor receptor tyrosine kinases. Cancer Chemother Pharmacol. 2013 Jul;72(1):53-64. doi: 10.1007/s00280-013-2168-z. Epub 2013 May 30. PMID 23719718
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx